CLINICAL TRIAL: NCT02985008
Title: SMart Angioplasty Research Team: A Multi-center, Open, REtrospective and Prospective Observational Study to Investigate Clinical oUtcomes and Efficacy of Left Ventricular Assist Device for Korean Patients With Cardiogenic Shock : RESCUE
Brief Title: Clinical Outcomes and Efficacy of Left Ventricular Assist Device for Korean Patients With Cardiogenic Shock
Acronym: SMART-RESCUE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jeong Hoon Yang (Other)
Responsible Party: Sponsor-Investigator, Jeong Hoon Yang, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: 2016-03-130
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Shock, Cardiogenic
Keywords: Shock, IVBP, ECMO, In hospital death
MeSH Terms: conditions — Shock, Cardiogenic; Shock

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospectively and prospectively enrolled patients with cardiogenic shock in domestic manifolds and investigated the current state of treatment and clinical features of cardiogenic shock in Koreans and identified the factors that could improve the prognosis and the use of IABP and ECMO And to investigate its therapeutic effect.

DETAILED DESCRIPTION:
1. The selection / exclusion criteria for persons with cardiogenic shock should be verified by medical records from January 1, 2014 before the approval date of each institution's clinical trial screening committee.
2. If a cardiogenic shock to the selection criteria is found in the emergency room, general ward, or intensive care unit of the participating institutions, enroll in this study and fill in the information according to the e-CRF.
3. After 1, 6 and 12 months, visit the hospital for examination and procedures. The person in charge of the examination or the delegate of the examiner may follow the person by telephone or an outpatient visit.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years old or older
2. ① Systolic blood pressure is less than 90mmHg for more than 30 minutes despite the fluid therapy, or Use of pressure boosting agents is necessary.

   ② Peripheral hypopnea (cold skin, urine less than 30 cc per hour, impaired consciousness, lactate ≥2.0 mmol / l) or a person with pulmonary edema.
3. Causes of cardiogenic shock include acute myocardial infarction (including in coronary intervention), cardiomyopathy, myocarditis, pulmonary embolism, refractory ventricular tachycardia, shock during coronary intervention.
4. Those voluntarily consenting to the medical records and the data necessary for the study during the entire study period.

Exclusion Criteria:

1. Other causes except for cardiogenic shock (low blood pressure, septic, obstructive shock)
2. Shock with cardiac arrest outside the hospital
3. People with allergic reactions to anticoagulants such as heparin.
4. Those who refused active treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total: 1,000
  * Cardiogenic shock group with inserted IABP, ECMO : 400
  * Cardiogenic shock group without inserted IABP, ECMO : 600
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
In hospital death | for 1 year

SECONDARY OUTCOMES:
Death in 28days | 28days
Death in 1 year | 1 year
Death, myocardial infarction, stroke, re-admission due to heart failure during follow-up. | 1 year
Number of days of intensive care unit Number of days of intensive care unit | 1 year
hospitalization days | 1 year
Lactate 24 hour clearance | 1 year
Successful removal of left ventricular assist device (IABP, ECMO) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Yang, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thiele H, Allam B, Chatellier G, Schuler G, Lafont A. Shock in acute myocardial infarction: the Cape Horn for trials? Eur Heart J. 2010 Aug;31(15):1828-35. doi: 10.1093/eurheartj/ehq220. Epub 2010 Jul 7. PMID 20610640
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, de Waha A, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Lauer B, Bohm M, Ebelt H, Schneider S, Werdan K, Schuler G; Intraaortic Balloon Pump in cardiogenic shock II (IABP-SHOCK II) trial investigators. Intra-aortic balloon counterpulsation in acute myocardial infarction complicated by cardiogenic shock (IABP-SHOCK II): final 12 month results of a randomised, open-label trial. Lancet. 2013 Nov 16;382(9905):1638-45. doi: 10.1016/S0140-6736(13)61783-3. Epub 2013 Sep 3. PMID 24011548
- [Background] Rousse N, Juthier F, Pincon C, Hysi I, Banfi C, Robin E, Fayad G, Jegou B, Prat A, Vincentelli A. ECMO as a bridge to decision: Recovery, VAD, or heart transplantation? Int J Cardiol. 2015;187:620-7. doi: 10.1016/j.ijcard.2015.03.283. Epub 2015 Mar 20. PMID 25863737
- [Background] Napp LC, Brehm M, Kuhn C, Schafer A, Bauersachs J. Heart against veno-arterial ECMO: Competition visualized. Int J Cardiol. 2015;187:164-5. doi: 10.1016/j.ijcard.2015.03.311. Epub 2015 Mar 21. No abstract available. PMID 25828345
- [Derived] Park IH, Kim CH, Jang WJ, Oh JH, Lee WS, Yang JH, Gwon HC. Sex-Specific Differences in Management and Outcomes of Cardiogenic Shock Patients With and Without Ischemic Cardiomyopathy. Korean Circ J. 2025 Sep;55(9):795-809. doi: 10.4070/kcj.2024.0440. Epub 2025 May 28. PMID 40537419
- [Derived] Kim O, Hong D, Choi KH, Lee JM, Park TK, Song YB, Hahn JY, Choi SH, Cho YH, Gwon HC, Yang JH. Sex Differences in Patients With Cardiogenic Shock Receiving Venoarterial Extracorporeal Membrane Oxygenation. Korean Circ J. 2025 Jun;55(6):541-551. doi: 10.4070/kcj.2024.0330. Epub 2025 Feb 10. PMID 40097285
- [Derived] Cha JH, Choi KH, Ahn CM, Yu CW, Park IH, Jang WJ, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD, Park TK, Lee JM, Song YB, Hahn JY, Choi SH, Gwon HC, Yang JH. Machine learning prediction of in-hospital mortality and external validation in patients with cardiogenic shock: the RESCUE score. Rev Esp Cardiol (Engl Ed). 2025 Aug;78(8):707-716. doi: 10.1016/j.rec.2025.01.003. Epub 2025 Jan 22. English, Spanish. PMID 39855461
- [Derived] Jung S, Jang WJ, Lee WS, Park IH, Oh JH, Yang JH, Gwon HC, Ahn CM, Yu CW, Kim HJ, Bae JW, Kwon SU, Lee HJ, Jeong JO, Park SD. Seasonal variation and prognosis in patients with acute myocardial infarction complicated by cardiogenic shock. Heliyon. 2024 Apr 24;10(9):e30078. doi: 10.1016/j.heliyon.2024.e30078. eCollection 2024 May 15. PMID 38720697
- [Derived] Hong D, Choi KH, Ahn CM, Yu CW, Park IH, Jang WJ, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD, Park TK, Lee JM, Song YB, Hahn JY, Choi SH, Gwon HC, Yang JH. Clinical significance of residual ischaemia in acute myocardial infarction complicated by cardiogenic shock undergoing venoarterial-extracorporeal membrane oxygenation. Eur Heart J Acute Cardiovasc Care. 2024 Jul 24;13(7):525-534. doi: 10.1093/ehjacc/zuae058. PMID 38701179
- [Derived] Jang WJ, Park IH, Oh JH, Choi KH, Song YB, Hahn JY, Choi SH, Gwon HC, Ahn CM, Yu CW, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD, Yang JH. Efficacy and safety of durable versus biodegradable polymer drug-eluting stents in patients with acute myocardial infarction complicated by cardiogenic shock. Sci Rep. 2024 Mar 15;14(1):6301. doi: 10.1038/s41598-024-56925-2. PMID 38491111
- [Derived] Jeong JH, Kook H, Lee SH, Joo HJ, Park JH, Hong SJ, Kim MN, Park SM, Jung JS, Yang JH, Gwon HC, Ahn CM, Jang WJ, Kim HJ, Bae JW, Kwon SU, Lee WS, Jeong JO, Park SD, Lim SH, Lee J, Lee J, Yu CW. Prediction of In-Hospital Mortality for Ischemic Cardiogenic Shock Requiring Venoarterial Extracorporeal Membrane Oxygenation. J Am Heart Assoc. 2024 Feb 20;13(4):e032701. doi: 10.1161/JAHA.123.032701. Epub 2024 Feb 16. PMID 38362865
- [Derived] Kim Y, Jang WJ, Park IH, Oh JH, Yang JH, Gwon HC, Ahn CM, Yu CW, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD. Prognostic effect of sex according to shock severity in patients with acute myocardial infarction complicated by cardiogenic shock. Hellenic J Cardiol. 2025 Mar-Apr;82:3-14. doi: 10.1016/j.hjc.2023.11.007. Epub 2023 Dec 10. PMID 38072307
- [Derived] Lee HH, Jang WJ, Ahn CM, Chun WJ, Oh JH, Park YH, Lee SJ, Hong SJ, Yang JH, Kim JS, Kim HC, Kim BK, Yu CW, Kim HJ, Bae JW, Ko YG, Choi D, Gwon HC, Hong MK, Jang Y. Association of Prophylactic Distal Perfusion Cannulation With Mortality in Patients Receiving Venoarterial Extracorporeal Membrane Oxygenation. Am J Cardiol. 2023 Nov 15;207:418-425. doi: 10.1016/j.amjcard.2023.07.149. Epub 2023 Oct 3. PMID 37797547
- [Derived] Choi KH, Yang JH, Park TK, Lee JM, Song YB, Hahn JY, Choi SH, Ahn CM, Yu CW, Park IH, Jang WJ, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD, Kang TS, Gwon HC. Culprit-Only Versus Immediate Multivessel Percutaneous Coronary Intervention in Patients With Acute Myocardial Infarction Complicating Advanced Cardiogenic Shock Requiring Venoarterial-Extracorporeal Membrane Oxygenation. J Am Heart Assoc. 2023 May 16;12(10):e029792. doi: 10.1161/JAHA.123.029792. Epub 2023 May 9. PMID 37158104
- [Derived] Park IH, Jang WJ, Oh JH, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Ahn CM, Yu CW, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD. Non-culprit left main coronary artery disease in acute myocardial infarction complicated by cardiogenic shock. PLoS One. 2023 Mar 30;18(3):e0276711. doi: 10.1371/journal.pone.0276711. eCollection 2023. PMID 36996239
- [Derived] Kwon W, Choi KH, Yang JH, Chung YJ, Park TK, Lee JM, Song YB, Hahn JY, Choi SH, Ahn CM, Yu CW, Park IH, Jang WJ, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD, Gwon HC. Efficacy of thrombus aspiration in cardiogenic shock complicating acute myocardial infarction and high thrombus burden. Rev Esp Cardiol (Engl Ed). 2023 Sep;76(9):719-728. doi: 10.1016/j.rec.2023.01.009. Epub 2023 Feb 4. English, Spanish. PMID 36746233
- [Derived] Kwon W, Lee SH, Yang JH, Choi KH, Park TK, Lee JM, Song YB, Hahn JY, Choi SH, Ahn CM, Ko YG, Yu CW, Jang WJ, Kim HJ, Kwon SU, Jeong JO, Park SD, Cho S, Bae JW, Gwon HC. Impact of the Obesity Paradox Between Sexes on In-Hospital Mortality in Cardiogenic Shock: A Retrospective Cohort Study. J Am Heart Assoc. 2022 Jun 7;11(11):e024143. doi: 10.1161/JAHA.121.024143. Epub 2022 Jun 6. PMID 35658518
- [Derived] Park IH, Yang JH, Jang WJ, Chun WJ, Oh JH, Park YH, Ko YG, Yu CW, Kim BS, Kim HJ, Lee HJ, Jeong JO, Gwon HC. Clinical significance of lactate clearance in patients with cardiogenic shock: results from the RESCUE registry. J Intensive Care. 2021 Oct 18;9(1):63. doi: 10.1186/s40560-021-00571-7. PMID 34663479
- [Derived] Jang WJ, Park IH, Yang JH, Chun WJ, Oh JH, Park YH, Ko YG, Yu CW, Kim HJ, Kim BS, Lee HJ, Jeong JO, Gwon HC. Association between polyvascular disease and clinical outcomes in patients with cardiogenic shock: Results from the RESCUE registry. Int J Cardiol. 2021 Sep 15;339:70-74. doi: 10.1016/j.ijcard.2021.07.008. Epub 2021 Jul 8. PMID 34246725
- [Derived] Seong SW, Jin G, Kim M, Ahn KT, Yang JH, Gwon HC, Ko YG, Yu CW, Chun WJ, Jang WJ, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Park SD, Cho SS, Ahn JH, Song PS, Jeong JO. Comparison of in-hospital outcomes of patients with vs. without ischaemic cardiomyopathy undergoing veno-arterial-extracorporeal membrane oxygenation. ESC Heart Fail. 2021 Aug;8(4):3308-3315. doi: 10.1002/ehf2.13481. Epub 2021 Jun 18. PMID 34145983
- [Derived] Yang JH, Choi KH, Ko YG, Ahn CM, Yu CW, Chun WJ, Jang WJ, Kim HJ, Kim BS, Bae JW, Lee SY, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD, Lim SH, Cho S, Park TK, Lee JM, Song YB, Hahn JY, Choi SH, Gwon HC. Clinical Characteristics and Predictors of In-Hospital Mortality in Patients With Cardiogenic Shock: Results From the RESCUE Registry. Circ Heart Fail. 2021 Jun;14(6):e008141. doi: 10.1161/CIRCHEARTFAILURE.120.008141. Epub 2021 Jun 15. PMID 34129366
- [Derived] Choi KH, Yang JH, Park TK, Lee JM, Song YB, Hahn JY, Choi SH, Ko YG, Yu CW, Chun WJ, Jang WJ, Kim HJ, Bae JW, Kwon SU, Lee HJ, Lee WS, Jeong JO, Park SD, Cho S, Gwon HC. Differential Prognostic Implications of Vasoactive Inotropic Score for Patients With Acute Myocardial Infarction Complicated by Cardiogenic Shock According to Use of Mechanical Circulatory Support. Crit Care Med. 2021 May 1;49(5):770-780. doi: 10.1097/CCM.0000000000004815. PMID 33590998
- [Derived] Lee HH, Hong SJ, Ahn CM, Yang JH, Gwon HC, Kim JS, Kim BK, Ko YG, Choi D, Hong MK, Jang Y. Clinical Implications of Thrombocytopenia at Cardiogenic Shock Presentation: Data from a Multicenter Registry. Yonsei Med J. 2020 Oct;61(10):851-859. doi: 10.3349/ymj.2020.61.10.851. PMID 32975059